CLINICAL TRIAL: NCT05892861
Title: The Effect of Multidomain Dietary Education in Type 2 Diabetic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Kaohsiung Normal University (Other)
Collaborators: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Ou Ling-Chun, Principal Investigator, National Kaohsiung Normal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 21-065-B
Record Dates: First submitted 2023-05-14; First posted 2023-06-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2023-06

CONDITIONS: Type2 Diabetes Mellitus; Cognitive Impairment, Mild
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- multi domain dietary education as cognitive stimulation (Experimental): video lifestyle education, board game, and 24-hour dietary recall record from 1st week to 10th week as cognitive stimulation.
  Interventions: Behavioral: cognitive stimulation
- usual clinical treatment (Experimental): usual treatment in clinic
  Interventions: Other: as usual care

INTERVENTIONS:
Behavioral: cognitive stimulation — video education, board games, and 24-hour dietary recall record
  Arms: multi domain dietary education as cognitive stimulation
Other: as usual care — history taking, explain data, and discuss how to control healthy condition
  Arms: usual clinical treatment

SUMMARY:
The goal of this clinical trial is to [learn about cognitive stimulation by multidomain dietary education including the dietary board game via LINE in non-dementic type 2 diabetic adults. The main questions it aims to answer are:

[Question 1: Could multi-domain dietary education as cognitive stimulation improve cognitive function?] [Question 2: Could multi-domain dietary education improve dietary control belief ?] [Question 3: Could multi-domain dietary education improve health behavior?] [Question 4]: Could multi-domain dietary education improve HbA1C, and lipid profile? Participants of experimental A group will receive a video about lifestyle education 5 minutes weekly for 3 weeks, a dietary board game 10 minutes weekly for 10 weeks, and a 24-hour dietary recall record 2 times weekly for 7 weeks. And participants of the experimental B group receive the usual clinical treatment. Then experimental A and Experimental B groups will cross over 12 weeks later.

Researchers will compare the effect of intervention between the experimental A group and the experimental B group.

DETAILED DESCRIPTION:
Cognitive function was measured by the Saint Louis University Mental State (SLUMS) score. And we exclude the dementia group according to the SLUMS definition (<21 if the participants graduated from senior high school or above, <20 if the education level below senior high school).

Experimental group A received 10-week curriculum from 1st week to 10th week, and receive d usual clinical care from 13th week to 22th week. Experimental B group received usual clinical care from 1st week to 10th week, and received 10-week curriculum from 13th week to 22th week.

ELIGIBILITY:
Inclusion Criteria:

* The onset age of Diabetes Mellitus is more than 20 years old
* Diagnosis of Diabetes according to past history including type 2 diabetes mellitus or drug history including oral anti-diabetic drugs

Exclusion Criteria:

* SLUMS meets the Dementia definition.
* HbA1C ≥ 10.0%
* Rejected our study.
* History of stroke.
* History of depression.
* History of psychiatric disease.
* Visual impairment.
* Hearing impairment.
* Can't understand the informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The change of cognitive function from baseline at 3 and 6 months | 12th week & 24 week
  Saint Louis University Mental State examination, the total score range is 0~30. Higher scores mean better change.

SECONDARY OUTCOMES:
The change of dietary control belief from baseline at 3 and 6 months | 12th week and 24th week
  12 questions by Linkert scale (4 questions about dietary mastery items and 8 questions about dietary perceived constraints items) about dietary control belief(the total score range is 12 to 60) Higher scores mean better change.

OTHER OUTCOMES:
The change of the awareness of complication and health behavior from baseline at 3 and 6 months | 12th week and 24th week
  8 questions about the complications of type 2 DM (stroke, blind, wood healing, amputation, CKD, CAD, hypoglycemia, and Dementia) by Linkert scale (the total score range is 8 to 40). Higher scores mean better change.
The change of HbA1C from baseline at 3 and 6 months | 12th week and 24th week
  biomedical data after phlebotomy (HbA1C in %), Higher scores mean worse change.
The change of total cholesterol from baseline at 3 and 6 months | 12th week and 24th week
  biomedical data after phlebotomy (total cholesterol in mg/dl). Higher scores mean worse change.
The change of triglyceride from baseline at 3 and 6 months | 12th week and 24th week
  biomedical data after phlebotomy (triglyceride in mg/dl). Higher scores mean worse change.
The change of low-density lipoprotein cholesterol from baseline at 3 and 6 months | 12th week and 24th week
  biomedical data after phlebotomy (low-density lipoprotein cholesterol in mg/dl). Higher scores mean worse change.
The change of high-density lipoprotein cholesterol from baseline at 3 and 6 months | 12th week and 24th week
  biomedical data after phlebotomy (high-density lipoprotein cholesterol in mg/dl). Higher scores mean worse change.
The change of health behavior awareness from baseline at 3 and 6 months | 12th week and 24th week
  9 questions about health behavior (body weight measurement, foot care, blood pressure measurement, drug adherence, diet adherence, calculation of intake amount by hand when eating, smoking habits, drinking habits, and exercise habits) by Linkert scale (total score range is 9 to 45). Higher scores mean better change.
The change of health behavior frequency per week from baseline at 3 and 6 months | 12th week and 24th week
  9 questions about health behavior (body weight measurement, foot care, blood pressure measurement, drug adherence, diet adherence, calculation of intake amount by hand when eating, smoking habits, drinking habits, and exercise habits) by Linkert scale (total score range is 9 to 45). Higher scores mean better change.

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Chun Ou, Principal Investigator — National Kaohsiung Normal University
Locations (1):
- Yong-Kang Clinic, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No